CLINICAL TRIAL: NCT03635086
Title: Observer Blinded, Randomised Study to Investigate Safety, Tolerability and Long-term Immunogenicity of Different Dose Regimens and Formulations of MV-CHIK in Healthy Volunteers
Brief Title: Safety, Tolerability and Long-term Immunogenicity of Different Formulations of a Chikungunya Vaccine (V184-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Themis Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V184-005; 2018-000211-25 (EudraCT Number); MV-CHIK-205 (Other: Themisbio)
Record Dates: First submitted 2018-07-24; First posted 2018-08-17 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Chikungunya Virus Infection
Keywords: Chikungunya fever
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A: Two MV-CHIK lyophilized low dose (Experimental): Participants received two vaccinations with MV-CHIK lyophilized formulation, low dose, on day 0 and day 28.
  Interventions: Biological: MV-CHIK lyophilised formulation, low dose
- Group B: Two MV-CHIK liquid frozen low dose (Experimental): Participants received two vaccinations with MV-CHIK liquid frozen low dose formulation on day 0 and day 28.
  Interventions: Biological: MV-CHIK liquid frozen formulation, low dose
- Group C: Two MV-CHIK liquid low dose stabilizing and protecting solution (SPS®) (Experimental): Participants received two vaccinations with MV-CHIK liquid low dose SPS® formulation on day 0 and day 28.
  Interventions: Biological: MV-CHIK SPS® formulation, low dose
- Group D: Two MV-CHIK liquid frozen high dose (Experimental): Participants received two vaccinations with MV-CHIK liquid frozen high dose formulation on day 0 and day 28.
  Interventions: Biological: MV-CHIK liquid frozen formulation, high dose
- Group E: One MV-CHIK liquid frozen high dose/placebo (Experimental): Participants received one vaccination with MV-CHIK liquid frozen high dose formulation on day 0 and placebo on day 28.
  Interventions: Biological: MV-CHIK liquid frozen formulation, high dose; Other: Placebo

INTERVENTIONS:
Biological: MV-CHIK lyophilised formulation, low dose — MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, lyophilized low dose (powder for suspension in water for intramuscular [IM] injection): 5x10^4 ±0.5 log tissue culture infectious dose 50 (TCID50)/dose.
  Arms: Group A: Two MV-CHIK lyophilized low dose
Biological: MV-CHIK liquid frozen formulation, low dose — MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, liquid frozen low dose (suspension for IM injection): 1x10^5 ±0.5 log TCID50/dose.
  Arms: Group B: Two MV-CHIK liquid frozen low dose
Biological: MV-CHIK SPS® formulation, low dose — MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, liquid SPS® low dose (suspension for IM injection): 1x10^5 ±0.5 log TCID50/dose.
  Arms: Group C: Two MV-CHIK liquid low dose stabilizing and protecting solution (SPS®)
Biological: MV-CHIK liquid frozen formulation, high dose — MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, liquid frozen high dose (suspension for IM injection): 1x10^6 ±0.5 log TCID50/dose.
  Arms: Group D: Two MV-CHIK liquid frozen high dose; Group E: One MV-CHIK liquid frozen high dose/placebo
Other: Placebo — Sterile physiological saline solution (0.9% sodium chloride [NaCl]), administered by IM injection.
  Arms: Group E: One MV-CHIK liquid frozen high dose/placebo

SUMMARY:
The purpose of this study is to investigate immunogenicity and safety of Measles Virus-Chikungunya (MV-CHIK) vaccine in different dose regimens, 28 days after one or two vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Is able to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the investigator and to comply with the requirements of the entire study
* Has a negative serum pregnancy test at screening (for female participants)
* Has a willingness not to become pregnant or to father a child during the entire study period by practicing reliable methods of contraception
* Has availability during the duration of the trial

Exclusion Criteria:

* Has participated in another clinical study (including exposure to an investigational medicinal product or device) within one month before the screening visit or planned concurrent participation in another clinical study before completion of the treatment period
* Has a history of immunodeficiency, known human immunodeficiency virus (HIV) infection or current hepatitis B/C infection
* Has a history of drug addiction including alcohol dependence within the last 2 years
* Has an inability or unwillingness to avoid intake of more than around 20 grams alcohol per day during 48 hours after each vaccination (equals roughly 0.5 liter beer or 0.25 liter of wine)
* Has had a vaccination within 4 weeks prior to first vaccination or planning to receive any non-study vaccine until end of treatment period
* Has had a prior receipt of any Chikungunya vaccine
* Has a history of moderate or severe arthritis or arthralgia within the past 3 months prior to screening
* Has had a recent infection within 1 week prior to screening
* Has made blood donations including plasma donations, 90 days prior to screening visit and anticipated blood, plasma, tissue, sperm or organ donation, throughout the study until end of treatment period
* Has clinically relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, hematological, endocrine, inflammatory, autoimmune or neurological diseases or clinically relevant abnormal laboratory values, that in the opinion of the investigator may interfere with the aim of the study
* Has a history of neoplastic disease (excluding non-melanoma skin cancer that was successfully treated) within the past 5 years or a history of any hematological malignancy
* Has behavioral, cognitive, or psychiatric condition that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Has a history of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the vaccine
* Has a history of anaphylaxis to drugs or other allergic reactions, which the investigator considers compromising the safety of the participant.
* Use of medication during 2 weeks before the first vaccination and throughout the study, which the investigator considers affecting the validity of the study, except hormonal contraception or hormonal replacement therapy in female participants.
* Use of immunosuppressive drugs like corticosteroids (excluding topical preparations) within 30 days prior to the first vaccination or anticipated use before completion of the treatment period
* Has receipt of blood products or immunoglobulins within 120 days prior to the screening visit or anticipated receipt of any blood product or immunoglobulin before completion of the treatment period
* Has pregnancy (positive pregnancy test at screening or during the treatment period) or lactation at screening, or planning to become pregnant during the treatment period
* Has unreliable contraception methods
* Is a person in a direct relationship with the sponsor, an investigator or other study team members. Direct dependent relationships include close relatives (i.e. children, parents, partner/spouse, siblings) as well as employees of the study site or the sponsor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ramsauer K, Schwameis M, Firbas C, Mullner M, Putnak RJ, Thomas SJ, Despres P, Tauber E, Jilma B, Tangy F. Immunogenicity, safety, and tolerability of a recombinant measles-virus-based chikungunya vaccine: a randomised, double-blind, placebo-controlled, active-comparator, first-in-man trial. Lancet Infect Dis. 2015 May;15(5):519-27. doi: 10.1016/S1473-3099(15)70043-5. Epub 2015 Mar 2. PMID 25739878

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After completion of screening procedures, participants will be randomized to one of five treatment groups (A, B, C, D or E).
Groups:
- Group A: Two Measles Virus-Chikungunya (MV-CHIK) Lyophilized Low Dose: Participants received two vaccinations (Day 0 and Day 28) with MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, lyophilized low dose (powder for suspension in water for intramuscular [IM] injection): 5x10^4 ±0.5 log tissue culture infectious dose 50 (TCID50)/dose.
- Group B: Two MV-CHIK Liquid Frozen Low Dose: Participants received two vaccinations (Day 0 and Day 28) with MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, liquid frozen low dose (suspension for IM injection): 1x10^5 ±0.5 log TCID50/dose.
- Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®): Participants received two vaccinations (Day 0 and Day 28) with MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, liquid SPS® low dose (suspension for IM injection): 1x10^5 ±0.5 log TCID50/dose.
- Group D: Two MV-CHIK Liquid Frozen High Dose: Participants received two vaccinations (Day 0 and Day 28) with MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, liquid frozen high dose (suspension for IM injection): 1x10^6 ±0.5 log TCID50/dose.
- Group E: One MV-CHIK Liquid Frozen High Dose: Participants received one vaccination (Day 0) with MV-CHIK a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, liquid frozen high dose (suspension for IM injection): 1x10^6 ±0.5 log TCID50/dose and placebo (Day 28), a sterile physiological saline solution (0.9% sodium chloride [NaCl]), administered by IM injection.
Period: Overall Study
Arm/Group | Group A: Two Measles Virus-Chikungunya (MV-CHIK) Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Started | 12 | 12 | 12 | 12 | 12
Completed | 11 | 11 | 11 | 12 | 12
Not Completed | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal of consent | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Two MV-CHIK Lyophilized Low Dose: Participants received two vaccinations (Day 0 and Day 28) with MV-CHIK, a live-attenuated recombinant measles vaccine expressing Chikungunya virus antigens, lyophilized low dose (powder for suspension in water for intramuscular [IM] injection): 5x10^4 ±0.5 log tissue culture infectious dose 50 (TCID50)/dose.
- Total: Total of all reporting groups
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (9.52) | 34.6 (11.79) | 39.0 (11.60) | 36.3 (9.62) | 36.8 (7.52) | 36.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 6 | 6 | 23
  Male | 9 | 8 | 8 | 6 | 6 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 12 | 12 | 12 | 12 | 60
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer of Anti-Chikungunya Antibodies as Measured by 50% Plaque Reduction Neutralization Test 28 Days After Last MV-CHIK Vaccination
Description: Participant serum was collected for determination of antibody responses by 50% plaque reduction neutralization test (PRNT50). Geometric Mean Titer (GMT) of functional antibodies as measured by PRNT50 were assessed. Geometric mean titers and GMT ratios were estimated by applying an analysis of variance (ANOVA) including the factor treatment group. This was done using log10 transformed data and taking the anti-log of the resulting point estimates for the least squares means, least squares means differences and the corresponding 2 sided 95% confidence intervals (CI). P-values were also provided to compare GMTs between treatment groups adjusted for multiple comparisons according to Tukey Kramer.
Time Frame: 28 days after last vaccination (Up to Day 56)
Population: The analysis population included all randomized participants who received at least one investigational medicinal product (IMP) administration and had no major protocol deviation that could have had an impact on their immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11 | 11 | 9 | 11 | 11
Titer | 21.0 [9.9 to 44.5] | 19.1 [9.0 to 40.5] | 13.6 [5.9 to 31.2] | 45.7 [21.6 to 97.0] | 8.9 [4.2 to 18.8]
Statistical Analysis 1: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; GMT ratios were estimated by applying an analysis of variance (ANOVA) including the factor treatment group. This was done using log10 transformed data and taking the anti-log of the resulting point estimates for the least squares means, least squares means differences and the corresponding 2-sided 95% confidence intervals (CI). P-values were also provided to compare GMTs between treatment groups adjusted for multiple comparisons according to Tukey-Kramer; Test type: Other; p = 0.9998, Tukey-Kramer; Geometric Mean Ratio Estimate = 1.1, 95% CI 2-sided [0.2 to 4.9]
Statistical Analysis 2: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); GMT ratios were estimated by applying an analysis of variance (ANOVA) including the factor treatment group. This was done using log10 transformed data and taking the anti-log of the resulting point estimates for the least squares means, least squares means differences and the corresponding 2-sided 95% confidence intervals (CI). P values were also provided to compare GMTs between treatment groups adjusted for multiple comparisons according to Tukey-Kramer; Test type: Other; p = 0.9345, Tukey-Kramer; Geometric Mean Ratio Estimate = 1.5, 95% CI 2-sided [0.3 to 7.5]
Statistical Analysis 3: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5836, Tukey-Kramer; Geometric Mean Ratio Estimate = 0.5, 95% CI 2-sided [0.1 to 2.1]
Statistical Analysis 4: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4844, Tukey-Kramer; Geometric Mean Ratio Estimate = 2.4, 95% CI 2-sided [0.5 to 10.6]
Statistical Analysis 5: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9725, Tukey-Kramer; Geometric Mean Ratio Estimate = 1.4, 95% CI 2-sided [0.3 to 6.8]
Statistical Analysis 6: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.4715, Tukey-Kramer; Geometric Mean Ratio Estimate = 0.4, 95% CI 2-sided [0.1 to 1.9]
Statistical Analysis 7: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5969, Tukey-Kramer; Geometric Mean Ratio Estimate = 2.2, 95% CI 2-sided [0.5 to 9.6]
Statistical Analysis 8: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2043, Tukey-Kramer; Geometric Mean Ratio Estimate = 0.3, 95% CI 2-sided [0.1 to 1.4]
Statistical Analysis 9: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9388, Tukey-Kramer; Geometric Mean Ratio Estimate = 1.5, 95% CI 2-sided [0.3 to 7.4]
Statistical Analysis 10: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0251, Tukey-Kramer; Geometric Mean Ratio Estimate = 5.2, 95% CI 2-sided [1.2 to 23.1]

2. Secondary Outcome: Percentage of Participants With Solicited and Unsolicited Adverse Events
Description: An adverse event (AE) includes any untoward medical occurrence in a participant to whom an IMP has been administered, not necessarily caused by or related to that product. An AE can therefore be any unfavourable or unintended sign, abnormal laboratory finding, symptom or disease temporally associated with the use of an IMP whether or not considered related to the IMP. The percentage of participants with solicited and unsolicited AEs was assessed.
Time Frame: Up to Day 56
Population: The analysis population included all participants who entered in the study and received at least one IMP administration. All analyses based on the safety population were carried out using the actual treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Percentage of Participants | 83.3 | 91.7 | 58.3 | 83.3 | 91.7

3. Secondary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event
Description: A serious adverse event (SAE) is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, and consists of a congenital anomaly, birth defect or other important medical events. As per the protocol, adverse events were analyzed per treatment group but were not assessed with respect to individual vaccinations.
Time Frame: Up to Day 56
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Geometric Mean Titer of Anti-Chikungunya Antibodies as Measured by PRNT50
Description: Participant serum was collected at each visit (Day 0, 28, 56, 182, and 365) for determination of antibody response by PRNT50. These results represent geometric mean titers (titers <10 were set to 5 for protocol-specified analysis).
Time Frame: Up to Day 365
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11 | 11 | 10 | 11 | 11
Titer
  Day 0 | 5.0 [3.0 to 8.2] | 8.6 [5.3 to 14.2] | 5.0 [3.0 to 8.4] | 5.0 [3.0 to 8.2] | 5.0 [3.0 to 8.2]
  Day 28 | 7.2 [3.9 to 13.2] | 14.0 [7.6 to 25.6] | 6.3 [3.4 to 11.9] | 11.3 [6.2 to 20.8] | 8.9 [4.8 to 16.2]
  Day 56: number analyzed (Participants) | 11 | 11 | 9 | 11 | 11
  Day 56 | 21.0 [10.1 to 43.7] | 19.1 [9.2 to 39.7] | 13.6 [6.0 to 30.5] | 45.7 [22.0 to 95.2] | 6.9 [3.3 to 14.3]
  Day 182 | 13.8 [7.0 to 27.2] | 18.2 [9.2 to 35.9] | 10.5 [5.1 to 21.5] | 11.8 [6.0 to 23.4] | 6.8 [3.4 to 13.5]
  Day 365: number analyzed (Participants) | 10 | 11 | 9 | 11 | 11
  Day 365 | 7.2 [3.9 to 13.6] | 11.8 [6.5 to 21.5] | 8.9 [4.6 to 17.2] | 8.3 [4.6 to 15.0] | 5.0 [2.8 to 9.1]
Statistical Analysis 1: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5263, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.2 to 1.6]
Statistical Analysis 2: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.4 to 2.8]
Statistical Analysis 3: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.4 to 2.7]
Statistical Analysis 4: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.4 to 2.7]
Statistical Analysis 5: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 0.5500, ANOVA; Geometric Mean Ratio Estimate = 1.7, 95% CI 2-sided [0.6 to 4.7]
Statistical Analysis 6: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 0.5263, ANOVA; Geometric Mean Ratio Estimate = 1.7, 95% CI 2-sided [0.6 to 4.6]
Statistical Analysis 7: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5263, ANOVA; Geometric Mean Ratio Estimate = 1.7, 95% CI 2-sided [0.6 to 4.6]
Statistical Analysis 8: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.4 to 2.8]
Statistical Analysis 9: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.4 to 2.8]
Statistical Analysis 10: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.4 to 2.7]
Statistical Analysis 11: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5321, ANOVA; Geometric Mean Ratio Estimate = 0.5, 95% CI 2-sided [0.2 to 1.7]
Statistical Analysis 12: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9983, ANOVA; Geometric Mean Ratio Estimate = 1.1, 95% CI 2-sided [0.3 to 3.9]
Statistical Analysis 13: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8234, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.2 to 2.1]
Statistical Analysis 14: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9882, ANOVA; Geometric Mean Ratio Estimate = 0.8, 95% CI 2-sided [0.2 to 2.7]
Statistical Analysis 15: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.3778, ANOVA; Geometric Mean Ratio Estimate = 2.2, 95% CI 2-sided [0.6 to 7.6]
Statistical Analysis 16: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9878, ANOVA; Geometric Mean Ratio Estimate = 1.2, 95% CI 2-sided [0.4 to 4.1]
Statistical Analysis 17: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8213, ANOVA; Geometric Mean Ratio Estimate = 1.6, 95% CI 2-sided [0.5 to 5.3]
Statistical Analysis 18: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.6716, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.2 to 1.9]
Statistical Analysis 19: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9380, ANOVA; Geometric Mean Ratio Estimate = 0.7, 95% CI 2-sided [0.2 to 2.5]
Statistical Analysis 20: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9777, ANOVA; Geometric Mean Ratio Estimate = 1.3, 95% CI 2-sided [0.4 to 4.3]
Statistical Analysis 21: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9997, ANOVA; Geometric Mean Ratio Estimate = 1.1, 95% CI 2-sided [0.3 to 4.7]
Statistical Analysis 22: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9287, ANOVA; Geometric Mean Ratio Estimate = 1.5, 95% CI 2-sided [0.3 to 7.2]
Statistical Analysis 23: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5598, ANOVA; Geometric Mean Ratio Estimate = 0.5, 95% CI 2-sided [0.1 to 2.0]
Statistical Analysis 24: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 0.2117, ANOVA; Geometric Mean Ratio Estimate = 3.0, 95% CI 2-sided [0.7 to 13.1]
Statistical Analysis 25: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9699, ANOVA; Geometric Mean Ratio Estimate = 1.4, 95% CI 2-sided [0.3 to 6.6]
Statistical Analysis 26: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.4460, ANOVA; Geometric Mean Ratio Estimate = 0.4, 95% CI 2-sided [0.1 to 1.8]
Statistical Analysis 27: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.2920, ANOVA; Geometric Mean Ratio Estimate = 2.8, 95% CI 2-sided [0.6 to 11.9]
Statistical Analysis 28: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.1840, ANOVA; Geometric Mean Ratio Estimate = 0.3, 95% CI 2-sided [0.1 to 1.4]
Statistical Analysis 29: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7229, ANOVA; Geometric Mean Ratio Estimate = 2.0, 95% CI 2-sided [0.4 to 9.2]
Statistical Analysis 30: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.0052, ANOVA; Geometric Mean Ratio Estimate = 6.6, 95% CI 2-sided [1.5 to 28.6]
Statistical Analysis 31: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9777, ANOVA; Geometric Mean Ratio Estimate = 0.8, 95% CI 2-sided [0.2 to 3.0]
Statistical Analysis 32: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9812, ANOVA; Geometric Mean Ratio Estimate = 1.3, 95% CI 2-sided [0.3 to 5.3]
Statistical Analysis 33: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9979, ANOVA; Geometric Mean Ratio Estimate = 1.2, 95% CI 2-sided [0.3 to 4.5]
Statistical Analysis 34: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5880, ANOVA; Geometric Mean Ratio Estimate = 2.0, 95% CI 2-sided [0.5 to 7.9]
Statistical Analysis 35: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7973, ANOVA; Geometric Mean Ratio Estimate = 1.7, 95% CI 2-sided [0.4 to 7.0]
Statistical Analysis 36: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8992, ANOVA; Geometric Mean Ratio Estimate = 1.5, 95% CI 2-sided [0.4 to 6.0]
Statistical Analysis 37: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.2602, ANOVA; Geometric Mean Ratio Estimate = 2.7, 95% CI 2-sided [0.7 to 10.4]
Statistical Analysis 38: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9991, ANOVA; Geometric Mean Ratio Estimate = 0.9, 95% CI 2-sided [0.2 to 3.6]
Statistical Analysis 39: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9028, ANOVA; Geometric Mean Ratio Estimate = 1.5, 95% CI 2-sided [0.4 to 6.2]
Statistical Analysis 40: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7761, ANOVA; Geometric Mean Ratio Estimate = 1.7, 95% CI 2-sided [0.4 to 6.8]
Statistical Analysis 41: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7833, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.2 to 2.1]
Statistical Analysis 42: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9915, ANOVA; Geometric Mean Ratio Estimate = 0.8, 95% CI 2-sided [0.2 to 2.9]
Statistical Analysis 43: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9980, ANOVA; Geometric Mean Ratio Estimate = 0.9, 95% CI 2-sided [0.3 to 3.0]
Statistical Analysis 44: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9090, ANOVA; Geometric Mean Ratio Estimate = 1.4, 95% CI 2-sided [0.4 to 4.9]
Statistical Analysis 45: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9651, ANOVA; Geometric Mean Ratio Estimate = 1.3, 95% CI 2-sided [0.4 to 4.7]
Statistical Analysis 46: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9112, ANOVA; Geometric Mean Ratio Estimate = 1.4, 95% CI 2-sided [0.4 to 4.7]
Statistical Analysis 47: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.2570, ANOVA; Geometric Mean Ratio Estimate = 2.4, 95% CI 2-sided [0.7 to 7.8]
Statistical Analysis 48: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9999, ANOVA; Geometric Mean Ratio Estimate = 1.1, 95% CI 2-sided [0.3 to 3.8]
Statistical Analysis 49: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.6953, ANOVA; Geometric Mean Ratio Estimate = 1.8, 95% CI 2-sided [0.5 to 6.2]
Statistical Analysis 50: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7523, ANOVA; Geometric Mean Ratio Estimate = 1.7, 95% CI 2-sided [0.5 to 5.4]

5. Secondary Outcome: Percentage of CD4+CD69+ Chikungunya Virus Specific T-Cells
Description: Cellular immunogenicity was determined by the evaluation of T cell immune response. Blood was collected for the isolation of peripheral blood mononuclear cells (PBMCs). PBMCs were isolated from whole blood to determine functional Interleukin 2 (IL-2)-producing T cells on day 0, 14, 28, 42, and 56 and in a subset of participants.
Time Frame: Up to Day 56
Population: The analysis population included a subset of all randomized participants who received at least one investigational medicinal product (IMP) administration and had no major protocol deviation that could have had an impact on their immune response. Based on the protocol, only participants in subset Treatment Group D (MV-CHIK liquid frozen high dose formulation) were analyzed for t-cell response.
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD4+CD69+ (Day 0) | 0.0194 (0.0446)
  CD4+CD69+ (Day 14) | 0.1430 (0.1589)
  CD4+CD69+ (Day 28) | 0.1077 (0.2060)
  CD4+CD69+ (Day 42) | 0.2050 (0.2316)
  CD4+CD69+ (Day 56) | 0.1935 (0.2036)

6. Secondary Outcome: Percentage of CD4+CD69+CD137+ Chikungunya Virus Specific T-Cells
Description: as for outcome 5
Time Frame: Up to Day 56
Population: The analysis population included a subset of all randomized participants who received at least one investigational medicinal product (IMP) administration and had no major protocol deviation that could have had an impact on their immune response. Based on the protocol, a subset of the participants in treatment group D (MV-CHIK liquid frozen high dose formulation) were analyzed for t-cell response.
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD4+CD69+CD137+ (Day 0) | 0.0061 (0.0112)
  CD4+CD69+CD137+ (Day 14) | 0.0174 (0.0313)
  CD4+CD69+CD137+ (Day 28) | 0.0120 (0.0168)
  CD4+CD69+CD137+ (Day 42) | 0.0317 (0.0438)
  CD4+CD69+CD137+ (Day 56) | 0.0393 (0.0476)

7. Secondary Outcome: Percentage of CD4+CD137+ Chikungunya Virus Specific T-Cells
Description: as for outcome 5
Time Frame: Up to Day 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD4+CD137+ (Day 0) | 0.0528 (0.0509)
  CD4+CD137+ (Day 14) | 0.1595 (0.2105)
  CD4+CD137+ (Day 28) | 0.1492 (0.0932)
  CD4+CD137+ (Day 42) | 0.3484 (0.3428)
  CD4+CD137+ (Day 56) | 0.3994 (0.2713)

8. Secondary Outcome: Percentage of CD4+CD69+OX40+ Chikungunya Virus Specific T-Cells
Description: as for outcome 5
Time Frame: Up to Day 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD4+CD69+OX40+ (Day 0) | 0.0033 (0.0048)
  CD4+CD69+OX40+ (Day 14) | 0.0265 (0.0522)
  CD4+CD69+OX40+ (Day 28) | 0.0095 (0.0070)
  CD4+CD69+OX40+ (Day 42) | 0.0267 (0.0408)
  CD4+CD69+OX40+ (Day 56) | 0.0337 (0.0386)

9. Secondary Outcome: Percentage of CD4+OX40+ Chikungunya Virus Specific T-Cells
Description: Cellular immunogenicity will be determined by the evaluation of T cell immune response. Blood was collected for the isolation of peripheral blood mononuclear cells (PBMCs). PBMCs were isolated from whole blood to determine functional Interleukin 2 (IL-2)-producing T cells on day 0, 14, 28, 42, and 56 and in a subset of subjects.
Time Frame: Up to Day 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD4+OX40+ (Day 0) | 0.0062 (0.0158)
  CD4+OX40+ (Day 14) | 0.0745 (0.1007)
  CD4+OX40+ (Day 28) | 0.0269 (0.0280)
  CD4+OX40+ (Day 42) | 0.0492 (0.1012)
  CD4+OX40+ (Day 56) | 0.0698 (0.0997)

10. Secondary Outcome: Percentage of CD8+CD69+ Chikungunya Virus Specific T-Cells
Description: as for outcome 5
Time Frame: Up to Day 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD8+CD69+ (Day 0) | 0.1919 (0.2329)
  CD8+CD69+ (Day 14) | 0.3319 (0.6046)
  CD8+CD69+ (Day 28) | 0.4242 (0.6330)
  CD8+CD69+ (Day 42) | 0.1961 (0.2496)
  CD8+CD69+ (Day 56) | 0.2375 (0.2902)

11. Secondary Outcome: Percentage of CD8+CD69+CD137+ Chikungunya Virus Specific T-Cells
Description: as for outcome 5
Time Frame: Up to Day 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD8+CD69+CD137+ (Day 0) | 0.0005 (0.0018)
  CD8+CD69+CD137+ (Day 14) | 0.0139 (0.0229)
  CD8+CD69+CD137+ (Day 28) | 0.0184 (0.0454)
  CD8+CD69+CD137+ (Day 42) | 0.0148 (0.0171)
  CD8+CD69+CD137+ (Day 56) | 0.0380 (0.0392)

12. Secondary Outcome: Percentage of CD8+CD137+ Chikungunya Virus Specific T-Cells
Description: as for outcome 5
Time Frame: Up to Day 56
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of t-cells
Arm/Group | Group D: Two MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11
Percentage of t-cells
  CD8+CD137+ (Day 0) | 0.0194 (0.0334)
  CD8+CD137+ (Day 14) | 0.0294 (0.0366)
  CD8+CD137+ (Day 28) | 0.0224 (0.0377)
  CD8+CD137+ (Day 42) | 0.0341 (0.0595)
  CD8+CD137+ (Day 56) | 0.0607 (0.0557)

13. Secondary Outcome: Geometric Mean Titer of Anti-Chikungunya Antibodies Determined by Enzyme Linked Immunosorbent Assay
Description: Participant serum was collected at each visit (Day 0, 28, 56, 182, and 365) for determination of Chikungunya antibody response by enzyme linked immunosorbent assay (ELISA). The analysis of variance GMT of Chikungunya-ELISA antibodies between treatment groups is summarized.
Time Frame: Up to Day 365
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11 | 11 | 10 | 11 | 11
Titer
  Day 0 | 7.4 (0.0) | 14.5 (3907.50) | 7.4 (0.0) | 7.4 (0.0) | 7.4 (0.0)
  Day 28 | 9.7 (46.83) | 17.8 (4009.38) | 8.1 (3.69) | 14.1 (28.47) | 13.1 (8.74)
  Day 56 | 54.3 (306.39) | 90.0 (4369.43) | 54.7 (112.29) | 171.4 (307.41) | 9.8 (7.69)
  Day 182 | 15.6 (112.90) | 26.9 (3304.35) | 16.3 (92.58) | 26.5 (17.36) | 8.1 (4.66)
  Day 365: number analyzed (Participants) | 10 | 11 | 9 | 11 | 11
  Day 365 | 11.9 (112.80) | 23.8 (3087.93) | 15.8 (75.39) | 18.9 (18.52) | 9.4 (10.01)
Statistical Analysis 1: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5263, ANOVA; Geometric Mean Ratio Estimate = 0.5, 95% CI 2-sided [0.1 to 1.7]
Statistical Analysis 2: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.3 to 3.5]
Statistical Analysis 3: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.3 to 3.4]
Statistical Analysis 4: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.3 to 3.4]
Statistical Analysis 5: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 0.5500, ANOVA; Geometric Mean Ratio Estimate = 2.0, 95% CI 2-sided [0.6 to 7.0]
Statistical Analysis 6: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 0.5263, ANOVA; Geometric Mean Ratio Estimate = 2.0, 95% CI 2-sided [0.6 to 6.7]
Statistical Analysis 7: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5263, ANOVA; Geometric Mean Ratio Estimate = 2.0, 95% CI 2-sided [0.6 to 6.7]
Statistical Analysis 8: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.3 to 3.5]
Statistical Analysis 9: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.3 to 3.5]
Statistical Analysis 10: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 0; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.3 to 3.4]
Statistical Analysis 11: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7708, ANOVA; Geometric Mean Ratio Estimate = 0.5, 95% CI 2-sided [0.1 to 2.4]
Statistical Analysis 12: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9966, ANOVA; Geometric Mean Ratio Estimate = 1.2, 95% CI 2-sided [0.3 to 5.4]
Statistical Analysis 13: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9503, ANOVA; Geometric Mean Ratio Estimate = 0.7, 95% CI 2-sided [0.2 to 3.0]
Statistical Analysis 14: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9791, ANOVA; Geometric Mean Ratio Estimate = 0.7, 95% CI 2-sided [0.2 to 3.2]
Statistical Analysis 15: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.5739, ANOVA; Geometric Mean Ratio Estimate = 2.2, 95% CI 2-sided [0.5 to 9.8]
Statistical Analysis 16: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9918, ANOVA; Geometric Mean Ratio Estimate = 1.3, 95% CI 2-sided [0.3 to 5.4]
Statistical Analysis 17: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9748, ANOVA; Geometric Mean Ratio Estimate = 1.4, 95% CI 2-sided [0.3 to 5.9]
Statistical Analysis 18: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8270, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.1 to 2.6]
Statistical Analysis 19: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8930, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.1 to 2.8]
Statistical Analysis 20: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 28; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9999, ANOVA; Geometric Mean Ratio Estimate = 1.1, 95% CI 2-sided [0.3 to 4.7]
Statistical Analysis 21: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9105, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.1 to 3.2]
Statistical Analysis 22: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.2 to 5.5]
Statistical Analysis 23: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.3047, ANOVA; Geometric Mean Ratio Estimate = 0.3, 95% CI 2-sided [0.1 to 1.7]
Statistical Analysis 24: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment; p = 0.0423, ANOVA; Geometric Mean Ratio Estimate = 5.5, 95% CI 2-sided [1.0 to 29.2]
Statistical Analysis 25: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9213, ANOVA; Geometric Mean Ratio Estimate = 1.6, 95% CI 2-sided [0.3 to 9.1]
Statistical Analysis 26: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8092, ANOVA; Geometric Mean Ratio Estimate = 0.5, 95% CI 2-sided [0.1 to 2.8]
Statistical Analysis 27: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.0040, ANOVA; Geometric Mean Ratio Estimate = 9.1, 95% CI 2-sided [1.7 to 48.5]
Statistical Analysis 28: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.3347, ANOVA; Geometric Mean Ratio Estimate = 0.3, 95% CI 2-sided [0.1 to 1.8]
Statistical Analysis 29: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.0488, ANOVA; Geometric Mean Ratio Estimate = 5.6, 95% CI 2-sided [1.0 to 30.7]
Statistical Analysis 30: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 56; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.0001, ANOVA; Geometric Mean Ratio Estimate = 17.4, 95% CI 2-sided [3.3 to 92.2]
Statistical Analysis 31: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8831, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.1 to 3.0]
Statistical Analysis 32: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.2 to 5.2]
Statistical Analysis 33: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.8916, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.1 to 3.1]
Statistical Analysis 34: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7940, ANOVA; Geometric Mean Ratio Estimate = 1.9, 95% CI 2-sided [0.4 to 9.9]
Statistical Analysis 35: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9169, ANOVA; Geometric Mean Ratio Estimate = 1.6, 95% CI 2-sided [0.3 to 8.9]
Statistical Analysis 36: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 1.0000, ANOVA; Geometric Mean Ratio Estimate = 1.0, 95% CI 2-sided [0.2 to 5.2]
Statistical Analysis 37: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.2563, ANOVA; Geometric Mean Ratio Estimate = 3.3, 95% CI 2-sided [0.6 to 17.1]
Statistical Analysis 38: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9237, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.1 to 3.3]
Statistical Analysis 39: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7708, ANOVA; Geometric Mean Ratio Estimate = 2.0, 95% CI 2-sided [0.4 to 10.8]
Statistical Analysis 40: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 182; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.2661, ANOVA; Geometric Mean Ratio Estimate = 3.3, 95% CI 2-sided [0.6 to 16.9]
Statistical Analysis 41: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group B: Two MV-CHIK Liquid Frozen Low Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7614, ANOVA; Geometric Mean Ratio Estimate = 0.5, 95% CI 2-sided [0.1 to 2.6]
Statistical Analysis 42: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9905, ANOVA; Geometric Mean Ratio Estimate = 0.8, 95% CI 2-sided [0.1 to 4.3]
Statistical Analysis 43: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9330, ANOVA; Geometric Mean Ratio Estimate = 0.6, 95% CI 2-sided [0.1 to 3.3]
Statistical Analysis 44: Comparison: Group A: Two MV-CHIK Lyophilized Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9945, ANOVA; Geometric Mean Ratio Estimate = 1.3, 95% CI 2-sided [0.2 to 6.7]
Statistical Analysis 45: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®); Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9599, ANOVA; Geometric Mean Ratio Estimate = 1.5, 95% CI 2-sided [0.3 to 8.4]
Statistical Analysis 46: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9942, ANOVA; Geometric Mean Ratio Estimate = 1.3, 95% CI 2-sided [0.2 to 6.4]
Statistical Analysis 47: Comparison: Group B: Two MV-CHIK Liquid Frozen Low Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.4932, ANOVA; Geometric Mean Ratio Estimate = 2.5, 95% CI 2-sided [0.5 to 12.9]
Statistical Analysis 48: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group D: Two MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9983, ANOVA; Geometric Mean Ratio Estimate = 0.8, 95% CI 2-sided [0.2 to 4.6]
Statistical Analysis 49: Comparison: Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.9112, ANOVA; Geometric Mean Ratio Estimate = 1.7, 95% CI 2-sided [0.3 to 9.3]
Statistical Analysis 50: Comparison: Group D: Two MV-CHIK Liquid Frozen High Dose vs Group E: One MV-CHIK Liquid Frozen High Dose; Day 365; Test type: Other — Analysis of variance (ANOVA) for GMT of Chikungunya-ELISA antibodies between treatment groups; p = 0.7431, ANOVA; Geometric Mean Ratio Estimate = 2.0, 95% CI 2-sided [0.4 to 10.2]

14. Secondary Outcome: Geometric Mean Titer of Anti-Measles Antibodies Determined by ELISA
Description: Participant serum was collected at each visit (Day 0, 28, and 56) for determination of antibody responses by ELISA.
Time Frame: Up to Day 56
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 11 | 11 | 10 | 11 | 11
Titer
  Day 0 | 711.6 (1764.77) | 482.1 (1009.40) | 750.2 (1580.90) | 731.0 (1612.98) | 888.4 (1560.14)
  Day 28 | 1250.8 (1629.35) | 1120.3 (849.01) | 1207.7 (1642.33) | 2246.4 (1515.40) | 2116.2 (1527.25)
  Day 56 | 1476.8 (1672.10) | 1158.6 (1019.59) | 1355.4 (1818.08) | 3009.80 (1355.67) | 2011.8 (1852.26)

15. Secondary Outcome: Number of Participants With Abnormal Laboratory Hematology Values Reported as an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Abnormal laboratory hematology value was any AE reported under the System Organ Class of Investigations that was related to an abnormal laboratory hematology value.
Time Frame: Up to Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 1 | 0 | 0 | 0 | 4

16. Secondary Outcome: Number of Participants With Abnormal Laboratory Chemistry Values Reported as an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Abnormal laboratory chemistry value was any AE reported under the System Organ Class of Investigations that was related to an abnormal laboratory chemistry value.
Time Frame: Up to Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants | 0 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events: Up to ~Day 56. All cause mortality: Up to ~Day 365.
Description: The analysis population included all participants who entered in the study and received at least one IMP administration. As per the protocol, adverse events were analyzed per treatment group but were not assessed with respect to individual vaccinations.
Arm/Group | Group A: Two MV-CHIK Lyophilized Low Dose | Group B: Two MV-CHIK Liquid Frozen Low Dose | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) | Group D: Two MV-CHIK Liquid Frozen High Dose | Group E: One MV-CHIK Liquid Frozen High Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12 | 7/12 | 10/12 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Two MV-CHIK Lyophilized Low Dose (N=12) | Group B: Two MV-CHIK Liquid Frozen Low Dose (N=12) | Group C: Two MV-CHIK Liquid Low Dose Stabilizing and Protecting Solution (SPS®) (N=12) | Group D: Two MV-CHIK Liquid Frozen High Dose (N=12) | Group E: One MV-CHIK Liquid Frozen High Dose (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (2)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (3)
Injection site pain (General disorders) | 2 (3) | 3 (5) | 3 (6) | 8 (15) | 7 (7)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (8) | 5 (7) | 5 (7) | 5 (7) | 5 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT03635086/Prot_SAP_000.pdf